CLINICAL TRIAL: NCT04455633
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of LX9211 in the Treatment of Diabetic Peripheral Neuropathic Pain
Brief Title: Efficacy, Safety, and PK of LX9211 in Participants With Diabetic Peripheral Neuropathic Pain
Acronym: RELIEF-DPN 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LX9211.1-201-DPN; LX9211.201 (Other: Lexicon Pharmaceuticals)
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Results first posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Diabetic Peripheral Neuropathy; Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Following a 2-week run-in period, participants were randomized to LX9211 matching placebo received as a single loading dose, orally, on Day 1, followed by maintenance doses of LX9211 matching placebo tablets, orally, once daily (QD) from Day 2 up to Week 6. Following completion of the 6-week treatment, all participants were followed for safety and received single oral tablet of LX9211 matching placebo, QD, for 5 weeks during the safety follow-up.
  Interventions: Drug: LX9211 Matching Placebo
- LX9211 100 mg/10 mg (Experimental): Following a 2-week run-in period, participants were randomized to receive a single loading dose of LX9211, 100 milligrams (mg), tablet, orally, on Day 1, followed by maintenance doses of LX9211 10 mg tablets, orally, QD from Day 2 up to Week 6. Following completion of the 6-week treatment, all participants were followed for safety and received single oral tablet of LX9211 matching placebo, QD, for 5 weeks during safety follow-up.
  Interventions: Drug: LX9211
- LX9211 200 mg/20 mg (Experimental): Following a 2-week run-in period, participants were randomized to receive a single loading dose of LX9211, 200 mg orally on Day 1, followed by maintenance doses of LX9211, 20 mg, orally, QD from Day 2 up to Week 6. Following completion of the 6-week treatment, all participants were followed for safety and received single oral tablet of LX9211 matching placebo, QD, for 5 weeks during safety follow-up.
  Interventions: Drug: LX9211

INTERVENTIONS:
Drug: LX9211 — Oral Tablets
  Arms: LX9211 100 mg/10 mg; LX9211 200 mg/20 mg
Drug: LX9211 Matching Placebo — Oral Tablets
  Arms: Placebo

SUMMARY:
Evaluation of the efficacy of a low and high dose of LX9211 compared to placebo in reducing pain related to diabetic peripheral neuropathy (DPNP) over an 11 week assessment period.

ELIGIBILITY:
Inclusion Criteria:

* Participant has given written informed consent to participate in the study in accordance with local regulations
* Adult male and female participants ≥18 years of age at the time of screening
* Body mass index ≥18.0 to ≤40.0 kg/m2 at Screening
* Diagnosis of diabetic peripheral neuropathic pain (DPNP) at Screening
* Pain from DPN present for at least 6 months
* Haemoglobin A1C ≤11% at screening
* Stable regimen for the treatment of type 1 diabetes mellitus (T1DM) or type 2 diabetes mellitus (T2DM) for ≥1 month prior to Screening

Exclusion Criteria:

* Presence of other painful conditions that may confound assessment or self-evaluation of DPNP
* History of major depressive episode, active, significant psychiatric disorders
* History of clinically significant drug or alcohol use disorder
* History of neurolytic or neurosurgical therapy for DPNP
* Use of opioid medications for management of DPNP within the 2 months prior to Screening Visit
* Use of non-steroidal anti-inflammatory drugs (NSAIDs) less than 2 weeks prior to the Screening Visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suma Gopinathan, PhD, Study Director — Lexicon Pharmaceuticals
Locations (42):
- United States (42):
  - Lexicon Investigational Site, Mobile, Alabama
  - Lexicon Investigational Site, Chandler, Arizona
  - Lexicon Investigational Site, Glendale, Arizona
  - Lexicon Investigational Site, Kingman, Arizona
  - Lexicon Investigational Site, Tucson, Arizona
  - Lexicon Investigational Site, Anaheim, California
  - Lexicon Investigational Site, Greenbrae, California
  - Lexicon Investigational Site, Los Angeles, California
  - Lexicon Investigational Site, North Hollywood, California
  - Lexicon Investigational Site, Sacramento, California
  - Lexicon Investigational Site, Tustin, California
  - Lexicon Investigational Site, Brandon, Florida
  - Lexicon Investigational Site, Fort Myers, Florida
  - Lexicon Investigational Site, Jacksonville, Florida
  - Lexicon Investigational Site, Lake City, Florida
  - Lexicon Investigational Site, New Port Richey, Florida
  - Lexicon Investigational Site, Ormond Beach, Florida
  - Lexicon Investigational Site, Winter Park, Florida
  - Lexicon Investigational Site, Macon, Georgia
  - Lexicon Investigational Site, Evansville, Indiana
  - Lexicon Investigational Site, Boston, Massachusetts
  - Lexicon Investigational Site, South Dartmouth, Massachusetts
  - Lexicon Investigational Site, Ann Arbor, Michigan
  - Lexicon Investigational Site, Dearborn, Michigan
  - Lexicon Investigational Site, Farmington Hills, Michigan
  - Lexicon Investigational Site, Sterling Heights, Michigan
  - Lexicon Investigational Site, Hazelwood, Missouri
  - Lexicon Investigational Site, Omaha, Nebraska
  - Lexicon Investigational Site, Berlin, New Jersey
  - Lexicon Investigational Site, Westfield, New York
  - Lexicon Investigational Site, Williamsville, New York
  - Lexicon Investigational Site, Asheville, North Carolina
  - Lexicon Investigational Site, Cary, North Carolina
  - Lexicon Investigational Site, Morehead City, North Carolina
  - Lexicon Investigational Site, Greenville, South Carolina
  - Lexicon Investigational Site, Austin, Texas
  - Lexicon Investigational Site, Dallas, Texas
  - Lexicon Investigational Site, Flower Mound, Texas
  - Lexicon Investigational Site, Houston, Texas
  - Lexicon Investigational Site, Pearland, Texas
  - Lexicon Investigational Site, Salt Lake City, Utah
  - Lexicon Investigational Site, Renton, Washington

REFERENCES:
- [Derived] Luo G, Chen L, Kostich WA, Hamman B, Allen J, Easton A, Bourin C, Gulianello M, Lippy J, Nara S, Maishal TK, Thiyagarajan K, Jalagam P, Pattipati SN, Dandapani K, Dokania M, Vattikundala P, Sharma V, Elavazhagan S, Verma MK, Das ML, Wagh S, Balakrishnan A, Johnson BM, Santone KS, Thalody G, Denton R, Saminathan H, Holenarsipur VK, Kumar A, Rao A, Putlur SP, Sarvasiddhi SK, Shankar G, Louis JV, Ramarao M, Conway CM, Li YW, Pieschl R, Tian Y, Hong Y, Ditta J, Mathur A, Li J, Smith D, Pawluczyk J, Sun D, Yip S, Wu DR, Vetrichelvan M, Gupta A, Wilson A, Gopinathan S, Wason S, Bristow L, Albright CF, Bronson JJ, Macor JE, Dzierba CD. Discovery of (S)-1-((2',6-Bis(difluoromethyl)-[2,4'-bipyridin]-5-yl)oxy)-2,4-dimethylpentan-2-amine (BMS-986176/LX-9211): A Highly Selective, CNS Penetrable, and Orally Active Adaptor Protein-2 Associated Kinase 1 Inhibitor in Clinical Trials for the Treatment of Neuropathic Pain. J Med Chem. 2022 Mar 24;65(6):4457-4480. doi: 10.1021/acs.jmedchem.1c02131. Epub 2022 Mar 8. PMID 35257579

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at multiple investigative sites in the United States from 03 Sep 2020 to 28 Jun 2022.
Pre-assignment Details: Participants with diagnosis of diabetic peripheral neuropathic pain were randomized in a 1:1:1 ratio to Placebo, LX9211 100 milligrams (mg)/10 mg and LX9211 200 mg/20 mg arm groups.
Groups:
- LX9211 100 mg/10 mg: Following a 2-week run-in period, participants were randomized to receive a single loading dose of LX9211, 100 mg tablet, orally, on Day 1, followed by maintenance doses of LX9211 10 mg tablet, orally, QD, from Day 2 up to Week 6. Following completion of the 6-week treatment, all participants were followed for safety and received single oral tablet of LX9211 matching placebo, QD, for 5 weeks during safety follow-up.
Period: Double-Blind Period (Up to Week 6)
Arm/Group | Placebo | LX9211 100 mg/10 mg | LX9211 200 mg/20 mg
Started (Randomized Participants.) | 107 | 106 | 106
Completed | 101 | 85 | 70
Not Completed | 6 | 21 | 36
Not completed — Adverse Event | 4 | 17 | 28
Not completed — Subject Choice Unrelated to Adverse Event/Serious Adverse Event | 2 | 2 | 6
Not completed — Other, not specified | 0 | 2 | 2
Period: Follow up Period (Weeks 7 to 11)
Arm/Group | Placebo | LX9211 100 mg/10 mg | LX9211 200 mg/20 mg
Started (Some of the participants who discontinued in double blind treatment period were also included in safety follow-up.) | 104 | 99 | 92
Completed | 103 | 99 | 92
Not Completed | 1 | 0 | 0
Not completed — Other, not specified | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The mITT population included all randomized participants who took at least 1 dose of study drug; participants were analyzed according to their randomized treatment.
Groups:
- Placebo: Following a 2-week run-in period, participants were randomized to LX9211 matching placebo received as a single loading dose, orally, on Day 1, followed by maintenance doses of LX9211 matching placebo tablets, orally, QD from Day 2 up to Week 6. Following completion of the 6-week treatment, all participants were followed for safety and received single oral tablet of LX9211 matching placebo, QD, for 5 weeks during the safety follow-up.
- Total: Total of all reporting groups
Arm/Group | Placebo | LX9211 100 mg/10 mg | LX9211 200 mg/20 mg | Total
Number analyzed (Participants) | 107 | 106 | 106 | 319
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (9.59) | 62.8 (9.26) | 61.8 (10.96) | 62.2 (9.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 48 | 43 | 132
  Male | 66 | 58 | 63 | 187
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 13 | 18 | 54
  Not Hispanic or Latino | 84 | 93 | 88 | 265
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 2
  Asian | 1 | 3 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 0 | 2
  Black or African American | 19 | 22 | 18 | 59
  White | 82 | 79 | 83 | 244
  Other | 3 | 0 | 4 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0
Average Daily Pain Score (ADPS) [Mean (Standard Deviation); unit: score on a scale] — Average Daily Pain Score (ADPS) is based on question 5 of Brief Pain Inventory (BPI)-short form for Diabetic Peripheral Neuropathy (BPI-DPN) and is assessed on an 11-point numerical rating scale. Participants were asked to rate their average pain over the past 24 hours, by answering the question 5 "Please rate your pain due to your diabetes by indicating the one number that best describes your pain on the average" on a scale of 0 to 10: 0=no pain, and 10=pain as bad as you can imagine. Higher ADPS scores indicate higher pain intensity. Population: The mITT population included all randomized participants who took at least 1 dose of study drug; participants were analyzed according to their randomized treatment. "Number analyzed" indicates number of participants with data available for analysis at Baseline.
  score on a scale
    number analyzed (Participants) | 106 | 106 | 104 | 316
    (all) | 6.54 (1.154) | 6.59 (1.091) | 6.53 (1.028) | 6.55 (1.089)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 6 in ADPS as Measured by the Numerical Rating Scale
Description: ADPS is based on question 5 of Brief Pain Inventory (BPI)-short form for Diabetic Peripheral Neuropathy (BPI-DPN) and is assessed on an 11-point numerical rating scale. Participants were asked to rate their average pain over the past 24 hours, by answering the question 5 "Please rate your pain due to your diabetes by indicating the one number that best describes your pain on the average." on a scale of 0 to 10: 0=no pain, and 10=pain as bad as you can imagine. Higher ADPS scores indicate higher pain intensity. Negative change from baseline indicates improvement.
Time Frame: Baseline (Week 2 of the Run-in period) to Week 6
Population: The modified intent to treat (mITT) population included all randomized participants who took at least 1 dose of study drug; participants were analyzed according to their randomized treatment. 'Overall number of participants analyzed' indicates the number of participants data available for the analysis of this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | LX9211 100 mg/10 mg | LX9211 200 mg/20 mg
Number analyzed (Participants) | 99 | 87 | 77
score on a scale | -0.72 [-1.08 to -0.36] | -1.39 [-1.77 to -1.01] | -1.27 [-1.66 to -0.88]
Statistical Analysis 1: Comparison: Placebo vs LX9211 100 mg/10 mg; Mixed model repeated measures (MMRM) model included fixed effects of treatment, visit, treatment-by-week interaction, the randomization stratum of Baseline pain severity (moderate, severe), and the Baseline ADPS score as a covariate; Test type: Superiority; p = 0.007, MMRM model; LS Mean Difference = -0.67, 95% CI 2-sided [-1.16 to -0.18], Standard Error of Mean 0.249
Statistical Analysis 2: Comparison: Placebo vs LX9211 200 mg/20 mg; MMRM model included fixed effects of treatment, visit, treatment-by-week interaction, the randomization stratum of Baseline pain severity (moderate, severe), and the Baseline ADPS score as a covariate; Test type: Superiority; p = 0.030, MMRM model; LS Mean Difference = -0.55, 95% CI 2-sided [-1.06 to -0.05], Standard Error of Mean 0.254

2. Secondary Outcome: Percentage of Participants With ≥30% Reduction in Pain Intensity in ADPS From Baseline to Week 6
Description: ADPS is based on question 5 of BPI-DPN and assessed on an 11-point numerical rating scale. Participants were asked to rate their average pain over the past 24 hours, by answering the question 5 "Please rate your pain due to your diabetes by indicating the one number that best describes your pain on the average." on a scale of 0 to 10 where 0 = No Pain and 10 = pain as bad as you can imagine. If % change from Baseline ≤ (-30) then participant was considered a Responder and if missing % change from Baseline or >(-30) participant is considered a Non-responder. Percentage of participants who were responders (who achieved ≥30% reduction in pain intensity in ADPS from Baseline to Week 6) are reported.
Time Frame: Baseline (Week 2 of the Run-in period) to Week 6
Population: The mITT population included all randomized participants who took at least 1 dose of study drug; participants were analyzed according to their randomized treatment. Missing observations at Week 6 are imputed as nonresponses.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | LX9211 100 mg/10 mg | LX9211 200 mg/20 mg
Number analyzed (Participants) | 107 | 106 | 106
percentage of participants | 17.8 | 27.4 | 17.0
Statistical Analysis 1: Comparison: Placebo vs LX9211 100 mg/10 mg; Percentage of responders were analyzed using the Cochran-Mantel-Haenszel (CMH) test stratified by the randomization factor of Baseline severity score (moderate, severe). The 95% confidence interval (CI) are calculated using the asymptotic Wald method. Missing observations at Week 6 are imputed as nonresponses; Test type: Superiority; p = 0.091, Cochran-Mantel-Haenszel; Difference in Percentage of Responders = 9.6, 95% CI 2-sided [-1.55 to 20.76]
Statistical Analysis 2: Comparison: Placebo vs LX9211 200 mg/20 mg; Percentage of responders were analyzed using the CMH test stratified by the randomization factor of Baseline severity score (moderate, severe). The 95% CI are calculated using the asymptotic Wald method. Missing observations at Week 6 are imputed as nonresponses; Test type: Superiority; p = 0.883, Cochran-Mantel-Haenszel; Difference in Percentage of Responders = -0.8, 95% CI 2-sided [-10.95 to 9.40]

3. Secondary Outcome: Percentage of Participants With ≥50% Reduction in Pain Intensity in ADPS From Baseline at Week 6
Description: ADPS is based on question 5 of BPI-DPN and assessed on an 11-point numerical rating scale. Participants were asked to rate their average pain over the past 24 hours, by answering the question 5 "Please rate your pain due to your diabetes by indicating the one number that best describes your pain on the average." on a scale of 0 to 10 where 0 = No Pain and 10 = pain as bad as you can imagine. If % change from Baseline ≤ (-50) then participant is considered a Responder and if missing % change from Baseline or >(-50) then participant is considered a Non-responder. Percentage of participants who were responders (who achieved ≥50% reduction in pain intensity in ADPS from Baseline to Week 6) are reported.
Time Frame: Baseline (Week 2 of the Run-in period) to Week 6
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | LX9211 100 mg/10 mg | LX9211 200 mg/20 mg
Number analyzed (Participants) | 107 | 106 | 106
percentage of participants | 10.3 | 15.1 | 9.4
Statistical Analysis 1: Comparison: Placebo vs LX9211 100 mg/10 mg; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.289, Cochran-Mantel-Haenszel; Difference in Percentage of Responders = 4.8, 95% CI 2-sided [-4.11 to 13.73]
Statistical Analysis 2: Comparison: Placebo vs LX9211 200 mg/20 mg; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.837, Cochran-Mantel-Haenszel; Difference in Percentage of Responders = -0.8, 95% CI 2-sided [-8.85 to 7.16]

4. Secondary Outcome: Change From Baseline to Week 6 in Severity of Pain and Interference of Pain With Sleep and Other Aspects of the Participant's Life Based on the BPI-DPN
Description: BPI-DPN: questionnaire that assesses severity of pain & its impact on functioning in participants with DPN. It consists of 4 questions that measure pain at its "worst,"least","average","now"(current pain) on 11-point numerical scale 0=no pain;10=worst pain.Score range:0-10 for each of these pain questions, higher scores=greater pain severity. Other 7 questions of BPI evaluate level of interference of pain on daily functioning (general activity,walking,work ability,mood,enjoyment of life,relations,sleep) on 11-point numerical scale, 0=does not interfere;10=completely interferes.Score range:0-10 for each of these intensity questions, higher scores=greater interference. Pain severity & pain interference factors are reported as separate categories. Average interference score= mean of 7 interference categories collected in Questions 9A-G, only if 50% (ie at least 4 of 7) of scores were non-missing. Negative change from baseline=improvement. Score range for average interference score: 0-70.
Time Frame: Baseline (Week 2 of the Run-in period) to Week 6
Population: The mITT population included all randomized participants who took at least 1 dose of study drug; participants were analyzed according to their randomized treatment. Overall number of participants analyzed' indicates the number of participants evaluable for the outcome measure analysis. Number analyzed indicates the number of participants evaluable for the outcome measure for the specified category.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | LX9211 100 mg/10 mg | LX9211 200 mg/20 mg
Number analyzed (Participants) | 89 | 77 | 86
score on a scale
  Pain at its Worst | -0.69 [-1.11 to -0.26] | -1.42 [-1.87 to -0.97] | -1.38 [-1.81 to -0.96]
  Pain at its Least | -0.69 [-1.13 to -0.26] | -1.43 [-1.89 to -0.98] | -1.38 [-1.81 to -0.95]
  Pain Right Now | -0.55 [-1.00 to -0.10] | -1.42 [-1.89 to -0.95] | -1.03 [-1.47 to -0.59]
  Interference Score Averaged Over Questions 9A - G | -0.74 [-1.17 to -0.30] | -1.00 [-1.46 to -0.53] | -0.97 [-1.41 to -0.53]
  General Activity | -0.77 [-1.25 to -0.28] | -0.96 [-1.48 to -0.44] | -0.82 [-1.31 to -0.33]
  Mood | -0.71 [-1.22 to -0.19] | -0.72 [-1.27 to -0.16] | -0.65 [-1.18 to -0.13]
  Walking Ability | -0.74 [-1.24 to -0.24] | -1.36 [-1.89 to -0.83] | -1.22 [-1.73 to -0.72]
  Normal Work | -1.01 [-1.50 to -0.53] | -1.07 [-1.58 to -0.55] | -1.05 [-1.54 to -0.56]
  Relations with Other People | -0.29 [-0.79 to 0.20] | 0.14 [-0.39 to 0.67] | -0.09 [-0.59 to 0.41]
  Sleep | -0.48 [-0.96 to -0.01] | -1.45 [-1.96 to -0.94] | -1.52 [-2.00 to -1.04]
  Enjoyment of Life | -1.03 [-1.53 to -0.52] | -1.05 [-1.59 to -0.50] | -1.13 [-1.64 to -0.61]
Statistical Analysis 1: Comparison: Placebo vs LX9211 100 mg/10 mg; Pain at its Worst: change from baseline was analyzed using MMRM model including fixed effects of treatment, visit, treatment-by-visit interaction, the randomization stratum of baseline pain severity (moderate, severe), and the baseline pain at its worst score as a covariate; Test type: Superiority; p = 0.014, MMRM model; LS Mean Difference = -0.73, 95% CI 2-sided [-1.32 to -0.15], Standard Error of Mean 0.298
Statistical Analysis 2: Comparison: Placebo vs LX9211 200 mg/20 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.017, MMRM model; LS Mean Difference = -0.70, 95% CI 2-sided [-1.27 to -0.13], Standard Error of Mean 0.290
Statistical Analysis 3: Comparison: Placebo vs LX9211 100 mg/10 mg; Pain at its Least: change from baseline was analyzed using MMRM model including fixed effects of treatment, visit, treatment-by-visit interaction, the randomization stratum of baseline pain severity (moderate, severe), and the baseline pain at its least score as a covariate; Test type: Superiority; p = 0.015, MMRM model; LS Mean Difference = -0.74, 95% CI 2-sided [-1.33 to -0.15], Standard Error of Mean 0.302
Statistical Analysis 4: Comparison: Placebo vs LX9211 200 mg/20 mg; [analysis description as in outcome 4, analysis 3]; Test type: Superiority; p = 0.020, MMRM model; LS Mean Difference = -0.69, 95% CI 2-sided [-1.27 to -0.11], Standard Error of Mean 0.294
Statistical Analysis 5: Comparison: Placebo vs LX9211 100 mg/10 mg; Pain Right Now: change from baseline was analyzed using MMRM model including fixed effects of treatment, visit, treatment-by-visit interaction, the randomization stratum of baseline pain severity (moderate, severe), and the baseline pain right now score as a covariate; Test type: Superiority; p = 0.005, MMRM model; LS Mean Difference = -0.87, 95% CI 2-sided [-1.48 to -0.27], Standard Error of Mean 0.309
Statistical Analysis 6: Comparison: Placebo vs LX9211 200 mg/20 mg; [analysis description as in outcome 4, analysis 5]; Test type: Superiority; p = 0.111, MMRM model; LS Mean Difference = -0.48, 95% CI 2-sided [-1.07 to 0.11], Standard Error of Mean 0.301
Statistical Analysis 7: Comparison: Placebo vs LX9211 100 mg/10 mg; Interference score averaged Over Questions 9A - G: change from baseline was analyzed using MMRM model including fixed effects of treatment, visit, treatment-by-visit interaction, the randomization stratum of baseline pain severity (moderate, severe), and the baseline pain interference score as a covariate; Test type: Superiority; p = 0.399, MMRM model; LS Mean Difference = -0.26, 95% CI 2-sided [-0.87 to 0.35], Standard Error of Mean 0.310
Statistical Analysis 8: Comparison: Placebo vs LX9211 200 mg/20 mg; [analysis description as in outcome 4, analysis 7]; Test type: Superiority; p = 0.441, MMRM model; LS Mean Difference = -0.23, 95% CI 2-sided [-0.83 to 0.36], Standard Error of Mean 0.302
Statistical Analysis 9: Comparison: Placebo vs LX9211 100 mg/10 mg; General Activity: change from baseline was analyzed using MMRM model including fixed effects of treatment, visit, treatment-by-visit interaction, the randomization stratum of baseline pain severity (moderate, severe), and the baseline general activity score as a covariate; Test type: Superiority; p = 0.575, MMRM model; LS Mean Difference = -0.19, 95% CI 2-sided [-0.87 to 0.49], Standard Error of Mean 0.346
Statistical Analysis 10: Comparison: Placebo vs LX9211 200 mg/20 mg; [analysis description as in outcome 4, analysis 9]; Test type: Superiority; p = 0.880, MMRM model; LS Mean Difference = -0.05, 95% CI 2-sided [-0.71 to 0.61], Standard Error of Mean 0.337
Statistical Analysis 11: Comparison: Placebo vs LX9211 100 mg/10 mg; Mood: change from baseline was analyzed using MMRM model including fixed effects of treatment, visit, treatment-by-visit interaction, the randomization stratum of baseline pain severity (moderate, severe), and the baseline mood score as a covariate; Test type: Superiority; p = 0.978, MMRM model; LS Mean Difference = -0.01, 95% CI 2-sided [-0.73 to 0.71], Standard Error of Mean 0.368
Statistical Analysis 12: Comparison: Placebo vs LX9211 200 mg/20 mg; [analysis description as in outcome 4, analysis 11]; Test type: Superiority; p = 0.877, MMRM model; LS Mean Difference = 0.06, 95% CI 2-sided [-0.65 to 0.76], Standard Error of Mean 0.358
Statistical Analysis 13: Comparison: Placebo vs LX9211 100 mg/10 mg; Walking Ability: change from baseline was analyzed using MMRM model including fixed effects of treatment, visit, treatment-by-visit interaction, the randomization stratum of baseline pain severity (moderate, severe), and the baseline walking ability score as a covariate; Test type: Superiority; p = 0.079, MMRM model; LS Mean Difference = -0.62, 95% CI 2-sided [-1.32 to 0.07], Standard Error of Mean 0.354
Statistical Analysis 14: Comparison: Placebo vs LX9211 200 mg/20 mg; [analysis description as in outcome 4, analysis 13]; Test type: Superiority; p = 0.163, MMRM model; LS Mean Difference = -0.48, 95% CI 2-sided [-1.16 to 0.20], Standard Error of Mean 0.345
Statistical Analysis 15: Comparison: Placebo vs LX9211 100 mg/10 mg; Normal Work: change from baseline was analyzed using MMRM model including fixed effects of treatment, visit, treatment-by-visit interaction, the randomization stratum of baseline pain severity (moderate, severe), and the baseline normal work score as a covariate; Test type: Superiority; p = 0.875, MMRM model; LS Mean Difference = -0.05, 95% CI 2-sided [-0.73 to 0.62], Standard Error of Mean 0.344
Statistical Analysis 16: Comparison: Placebo vs LX9211 200 mg/20 mg; [analysis description as in outcome 4, analysis 15]; Test type: Superiority; p = 0.914, MMRM model; LS Mean Difference = -0.04, 95% CI 2-sided [-0.69 to 0.62], Standard Error of Mean 0.335
Statistical Analysis 17: Comparison: Placebo vs LX9211 100 mg/10 mg; Relations with Other People: change from baseline was analyzed using MMRM model including fixed effects of treatment, visit, treatment-by-visit interaction, the randomization stratum of baseline pain severity (moderate, severe), and the baseline relations with other people score as a covariate; Test type: Superiority; p = 0.219, MMRM model; LS Mean Difference = 0.43, 95% CI 2-sided [-0.26 to 1.12], Standard Error of Mean 0.351
Statistical Analysis 18: Comparison: Placebo vs LX9211 200 mg/20 mg; [analysis description as in outcome 4, analysis 17]; Test type: Superiority; p = 0.551, MMRM model; LS Mean Difference = 0.20, 95% CI 2-sided [-0.47 to 0.87], Standard Error of Mean 0.341
Statistical Analysis 19: Comparison: Placebo vs LX9211 100 mg/10 mg; Sleep: change from baseline was analyzed using MMRM model including fixed effects of treatment, visit, treatment-by-visit interaction, the randomization stratum of baseline pain severity (moderate, severe), and the baseline sleep score as a covariate; Test type: Superiority; p = 0.005, MMRM model; LS Mean Difference = -0.96, 95% CI 2-sided [-1.63 to -0.30], Standard Error of Mean 0.339
Statistical Analysis 20: Comparison: Placebo vs LX9211 200 mg/20 mg; [analysis description as in outcome 4, analysis 19]; Test type: Superiority; p = 0.002, MMRM model; LS Mean Difference = -1.04, 95% CI 2-sided [-1.68 to -0.39], Standard Error of Mean 0.329
Statistical Analysis 21: Comparison: Placebo vs LX9211 100 mg/10 mg; Enjoyment of Life: change from baseline was analyzed using MMRM model including fixed effects of treatment, visit, treatment-by-visit interaction, the randomization stratum of baseline pain severity (moderate, severe), and the baseline enjoyment of life score as a covariate; Test type: Superiority; p = 0.955, MMRM model; LS Mean Difference = -0.02, 95% CI 2-sided [-0.73 to 0.69], Standard Error of Mean 0.361
Statistical Analysis 22: Comparison: Placebo vs LX9211 200 mg/20 mg; [analysis description as in outcome 4, analysis 21]; Test type: Superiority; p = 0.777, MMRM model; LS Mean Difference = -0.10, 95% CI 2-sided [-0.79 to 0.59], Standard Error of Mean 0.351

5. Secondary Outcome: Percentage of Participants Discontinuing Treatment Due to Lack of Efficacy
Description: Lack of efficacy was defined as an increase of 30% from baseline in ADPS based on question 5 of the BPI-DPN. Baseline was defined as the average of the Week 2 Run-in period data collected by participants in the daily pain diary of BPI-DPN. ADPS is based on question 5 of BPI-DPN and assessed on an 11-point numerical rating scale where 0 = No Pain to 10 = pain as bad as you can imagine, higher score indicates higher pain intensity.
Time Frame: Baseline (Week 2 of the Run-in period) to Week 6
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | LX9211 100 mg/10 mg | LX9211 200 mg/20 mg
Number analyzed (Participants) | 107 | 106 | 106
percentage of participants | 0 | 0 | 0

6. Secondary Outcome: Patient Global Impression of Change (PGIC) Scale Score at Week 6
Description: PGIC is a 7-point rating scale that assesses participant's belief about the overall improvement experienced after the end of treatment, where 1= very much improved to 7 = very much worse. Higher score indicates worsening.
Time Frame: Baseline (Week 2 of the Run-in period) to Week 6
Population: The mITT population included all randomized participants who took at least 1 dose of study drug; participants were analyzed according to their randomized treatment. Overall number of participants analyzed indicates the number of participants evaluable for the analysis of the outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | LX9211 100 mg/10 mg | LX9211 200 mg/20 mg
Number analyzed (Participants) | 103 | 99 | 94
score on a scale | 3.28 [3.04 to 3.52] | 2.93 [2.69 to 3.17] | 3.13 [2.88 to 3.38]
Statistical Analysis 1: Comparison: Placebo vs LX9211 100 mg/10 mg; Analysis of variance (ANOVA) model was used for the analysis with treatment and the randomization stratum of baseline pain severity (moderate, severe) as fixed covariates; Test type: Superiority; p = 0.031, ANOVA; LS Mean Difference = -0.35, 95% CI 2-sided [-0.67 to -0.03], Standard Error of Mean 0.163
Statistical Analysis 2: Comparison: Placebo vs LX9211 200 mg/20 mg; ANOVA model was used for the analysis with treatment and the randomization stratum of baseline pain severity (moderate, severe) as fixed covariates; Test type: Superiority; p = 0.351, ANOVA; LS Mean Difference = -0.15, 95% CI 2-sided [-0.48 to 0.17], Standard Error of Mean 0.165

7. Secondary Outcome: Time to Loss of Efficacy From Week 6 to Week 11 Among Participants Achieving a ≥30% Reduction in Pain Intensity at Week 6
Description: For participants who achieved ≥30% reduction in ADPS based on Question 5 of the BPI-DPN at Week 6, the time to loss of efficacy was defined as the time from the date of Week 6 visit to the date of termination of safety follow-up due to lack of efficacy. ADPS is based on question 5 of BPI-DPN and assessed on an 11-point numerical rating scale where, 0 = No Pain to 10 = pain as bad as you can imagine.
Time Frame: Weeks 6 to 11
Population: The mITT population included all randomized participants who took at least 1 dose of study drug; participants were analyzed according to their randomized treatment. Participants who had ≥30% Reduction in Pain Intensity in ADPS at Week 6 were analyzed for this outcome measure.
Measure: Median (Full Range); unit: weeks
Arm/Group | Placebo | LX9211 100 mg/10 mg | LX9211 200 mg/20 mg
Number analyzed (Participants) | 11 | 16 | 10
weeks | NA [NA to NA] — As none of the participants discontinued due to loss of efficacy during Weeks 6 to 11, median and full range could not be estimated. | NA [NA to NA] — As none of the participants discontinued due to loss of efficacy during Weeks 6 to 11, median and full range could not be estimated. | NA [NA to NA] — As none of the participants discontinued due to loss of efficacy during Weeks 6 to 11, median and full range could not be estimated.

8. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Adverse Events (AE) is defined as any sign, symptom, or diagnosis/disease that is unfavorable or unintended, that is new, or if pre-existing, worsens in participants administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. Treatment-emergent AEs are defined as any AEs that occur or worsen after the first dose of study medication.
Time Frame: First dose of study drug after randomization up to the end of study (up to Week 11)
Population: The safety population included those participants who took at least 1 dose of study drug during the double-blind treatment period. AEs were collected and reported for treatment period and safety follow up period separately.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo (Double-blind Treatment Period): Following a 2-week single-blind Run-in period, participants were randomized to receive a single loading dose of LX9211 matching placebo tablet, orally, on Day 1 and maintenance doses, orally, once daily from Day 2 to Week 6 during the 6-week double-blind treatment period.
- LX9211 100 mg/10 mg (Double-blind Treatment Period): Following a 2-week Single-blind Run-in period, participants were randomized to receive a single loading dose of 100 mg tablet, orally, on Day 1 and maintenance doses of 10 mg, orally, once daily from Day 2 to Week 6 during the 6-week double-blind treatment period.
- LX9211 200 mg/20 mg (Double-blind Treatment Period): Following a 2-week Single-blind Run-in period, participants were randomized to receive a single loading dose of 200 mg tablet, orally, on Day 1 and maintenance doses of 20 mg, orally, once daily from Day 2 to Week 6 during the 6-week double-blind treatment period.
- Placebo (Single-blind Follow-up Period); LX9211 100 mg/10 mg (Single-blind Follow-up Period); LX9211 200 mg/20 mg Single-blind Follow-up Period): Following completion of the 6-week double-blind treatment period, all participants entered the 5-week single-blind follow-up period and received a daily dose of LX9211 matching placebo tablet, orally.
Arm/Group | Placebo (Double-blind Treatment Period) | LX9211 100 mg/10 mg (Double-blind Treatment Period) | LX9211 200 mg/20 mg (Double-blind Treatment Period) | Placebo (Single-blind Follow-up Period) | LX9211 100 mg/10 mg (Single-blind Follow-up Period) | LX9211 200 mg/20 mg Single-blind Follow-up Period)
Number analyzed (Participants) | 107 | 106 | 106 | 104 | 99 | 92
Participants | 32 | 57 | 54 | 15 | 21 | 18

ADVERSE EVENTS:
Time Frame: First dose of study drug after randomization up to the end of study (up to Week 11)
Description: The safety population included those participants who took at least 1 dose of study drug during the double-blind treatment period. Adverse events reported occurred at a frequency >=5% in any treatment group. AEs were collected and reported for treatment period and safety follow up period separately.
Arm/Group | Placebo (Double-blind Treatment Period) | LX9211 100 mg/10 mg (Double-blind Treatment Period) | LX9211 200 mg/20 mg (Double-blind Treatment Period) | Placebo (Single-blind Follow-up Period) | LX9211 100 mg/10 mg (Single-blind Follow-up Period) | LX9211 200 mg/20 mg Single-blind Follow-up Period)
All-Cause Mortality (participants affected / at risk) | 1/107 | 0/106 | 1/106 | 0/104 | 0/99 | 0/92
Serious Adverse Events (participants affected / at risk) | 1/107 | 0/106 | 2/106 | 1/104 | 1/99 | 1/92
Other Adverse Events (participants affected / at risk) | 9/107 | 39/106 | 44/106 | 4/104 | 2/99 | 6/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Double-blind Treatment Period) (N=107) | LX9211 100 mg/10 mg (Double-blind Treatment Period) (N=106) | LX9211 200 mg/20 mg (Double-blind Treatment Period) (N=106) | Placebo (Single-blind Follow-up Period) (N=104) | LX9211 100 mg/10 mg (Single-blind Follow-up Period) (N=99) | LX9211 200 mg/20 mg Single-blind Follow-up Period) (N=92)
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Coronavirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Double-blind Treatment Period) (N=107) | LX9211 100 mg/10 mg (Double-blind Treatment Period) (N=106) | LX9211 200 mg/20 mg (Double-blind Treatment Period) (N=106) | Placebo (Single-blind Follow-up Period) (N=104) | LX9211 100 mg/10 mg (Single-blind Follow-up Period) (N=99) | LX9211 200 mg/20 mg Single-blind Follow-up Period) (N=92)
Dizziness (Nervous system disorders) | 2 | 16 | 29 | 2 | 1 | 1
Headache (Nervous system disorders) | 4 | 9 | 10 | 2 | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 6 | 5 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 7 | 2 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 9 | 12 | 1 | 0 | 3
Constipation (Gastrointestinal disorders) | 3 | 4 | 8 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2 | 7 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution must provide any proposed publication or presentation to Sponsor for Sponsor's review, comment and approval at least thirty (30) days prior to the proposed submission for publication date or the proposed presentation date. Sponsor shall have the right to have deleted from the final version of the publication any confidential information, proprietary information, or patentable participant matter.

DOCUMENTS (2):
  • Study Protocol (2021-09-09): https://cdn.clinicaltrials.gov/large-docs/33/NCT04455633/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-07): https://cdn.clinicaltrials.gov/large-docs/33/NCT04455633/SAP_001.pdf